CLINICAL TRIAL: NCT05574101
Title: A Phase II, Multicenter, Single-Arm Clinical Trial of Radiotherapy and CeMiPlimAb: Rwlc ImmunoTherapy for Locally Advanced, Unresectable Cutaneous Squamous Cell Carcinoma: RAMPART
Brief Title: A Study of Radiation Therapy and Cemiplimab for People With Skin Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-090
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Skin Cancer; Squamous Cell Carcinoma; Locally Advanced Squamous Cell Carcinoma; Locally Advanced Squamous Cell Carcinoma of the Skin; Locally Advanced Cutaneous Squamous Cell Carcinoma; Locally Advanced Skin Squamous Cell Carcinoma
Keywords: Skin cancer; squamous cell carcinoma; locally advanced squamous cell carcinoma; Cutaneous Squamous Cell Carcinoma; Locally Advanced Squamous Cell Carcinoma of the Skin; Locally Advanced Cutaneous Squamous Cell Carcinoma; Locally Advanced Skin Squamous Cell Carcinoma; cemiplimab; RAMPART; 22-090; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Skin Neoplasms; Carcinoma, Squamous Cell | interventions — cemiplimab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with locally advanced, unresectable cutaneous squamous cell carcinoma/CSCC (Experimental): Participants have locally advanced, unresectable cutaneous squamous cell carcinoma/CSCC
  Interventions: Drug: Cemiplimab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cemiplimab — Participants will undergo baseline imaging, followed by two doses of neoadjuvant cemiplimab at a dose of 350 mg intravenously over 30 minutes every 3 weeks (+/-3 days). Then, participants will receive concurrent cemiplimab 350 mg intravenously over 30 minutes every 3 weeks (+/-3 days) concurrently with RT to 70 Gy in 35 fractions over 7 weeks. Thereafter, participants will receive 38 weeks of cemiplimab 350 mg intravenously over 30 minutes every 3 weeks (+/-3 days) for a cumulative total of 12 months of cemiplimab.
Radiation: Radiotherapy — Participants will receive radiotherapy to 70 Gy in 35 fractions over 7 weeks concurrently with cemiplimab

SUMMARY:
The purpose of the study is to see if the combination of radiation therapy and cemiplimab immunotherapy is an effective treatment for people with locally advanced, unresectable CSCC.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven cutaneous squamous cell carcinoma which is locally advanced

  * Mixed histology tumors that are predominantly squamous cell carcinoma are eligible
  * Locally advanced primary tumor is T3-T4 and/or N+ by AJCC and/or UICC 8th edition clinical criteria
* T3-T4 primary tumor characteristics noted below:

  * Non-eyelid tumor >4 cm in maximum dimension or with bone erosion or invasion, perineural invasion of nerve 0.1 mm or larger, or invasion beyond subcutaneous fat or >6 mm from granular layer of adjacent normal epidermis
  * Eyelid tumor >2 cm or invading adjacent ocular, orbital or facial structures
* ≥18 years old
* Unresectable or medically inoperable according to local multidisciplinary consensus for reasons such as:

  * Tumor or regional lymph node metastases that has recurred despite ≥2 prior surgical procedures, with another curative resection unlikely
  * Tumor or nodal disease with significant local invasion that precludes complete resection
  * Tumor or nodal disease in anatomically challenging area where surgery may result in significant disfigurement or dysfunction (amputation of nose, ear, eye, digit, limb, etc)
  * Medical contraindication to surgery
  * Patient refusal of surgery due to anticipate morbidity
* ECOG ≤2
* Adequate bone marrow and metabolic function (by blood tests)

  * Total bilirubin ≤1.5 x upper limit of normal
  * Aspirate aminotransferase (AST) ≤3 x upper limit of normal
  * Alanine aminotransferase (ALT) ≤3 x upper limit of normal
  * Alkaline phosphatase ≤2.5 x upper limit of normal
  * Serum creatinine ≤1.5 x upper limit of normal or estimated creatinine clearance >30 mL/min according to Cockcroft-Gault formula
  * Hemoglobin >9 g/dL
  * Absolute neutrophil count ≥1.5 x10^9/L
  * Platelet count ≥75 x10^9/L
* Able to provide informed consent
* Acceptable candidate for curative intent radiotherapy and Cemiplimab immunotherapy, in opinion of radiation and medical oncologist, respectively
* Life expectancy >18 months

Exclusion Criteria:

* Primary tumor originating on the mucosal (non-hair bearing) lip or nose, anogenital (penis, scrotum, vulva, perianal) area
* Iatrogenic immunosuppression (>prednisone 10 mg/day or equivalent within 14 days of initiation of treatment)
* Women of child bearing potential unwilling or unable to use effective contraception while receiving treatment with cemiplimab and for 4 months thereafter
* Distant metastases
* Clinically significant autoimmune disease that requires iatrogenic immunosuppression

  o For example, severe rheumatoid arthritis requiring disease modifying antirheumatic drugs, such as methotrexate
* Current or previous hematopoietic malignancy (leukemia, lymphoma)
* Prior allogeneic transplant of solid organ or bone marrow
* Concurrent malignancies with >10% risk of metastasis or death within 2 years
* Prior aPD1 immunotherapy or PI3Kδ inhibitor use
* Prior radiotherapy for the cutaneous squamous cell carcinoma requiring treatment
* Other ongoing cancer therapy

  o Adjuvant endocrine therapy is permitted for patients with prostate or breast cancer
* Uncontrolled HIV or infectious hepatitis (viral load detectable in patient with known infection)
* Pregnancy or breastfeeding
* Comorbid or diagnostic abnormalities within the last year that would interfere with interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2026-10-06 (Estimated); Study Completion 2026-10-06 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | 18 months
  The primary endpoint for this study is disease free survival at 18 months (week 78 +/- 3 weeks) after starting cemiplimab.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Barker, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (13):
- United States (13):
  - University of Colorado (Data Collection Only), Aurora, Colorado
  - Moffitt Cancer Center (Data Collection Only), Tampa, Florida
  - Memorial Sloan Kettering Cancer Center at Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Rockville Centre, New York
  - Cleveland Clinic (Data Collection Only), Cleveland, Ohio
  - Fox Chase Cancer Center (Data Collection Only), Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Washington (Data Collection Only), Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org